CLINICAL TRIAL: NCT03103035
Title: Enhancing Knowledge Translation in Nutrition Through a Healthy Eating Blog: A Mixed Methods Feasibility Study
Brief Title: Enhancing Knowledge Translation in Nutrition Through a Healthy Eating Blog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-084 A-2 / 16-06-2015
Record Dates: First submitted 2015-04-08; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposition to a healthy eating blog (Experimental): Participants randomised to this arm are exposed to one blog post each week for a period of 6 months.
  Interventions: Other: Blog
- No exposition to a healthy eating blog (No Intervention): Participants randomised to this arm do not have exposure to the blog.

INTERVENTIONS:
Other: Blog — Participants randomised to the experimental group are exposed to one blog post each week for a period of 6 months. Blog posts focus on the improvement of fruits and vegetables consumption targeting four main determinants of the behavior: (1) knowledge; (2) attitude; (3) self-efficacy; and (4) motivation/goals. Each post included a step-by-step recipe developed by the research team and featuring fruits and vegetables. Recipes were described textually and also using pictures and/or video. Twenty-six posts were created over the six-month intervention.
  Arms: Exposition to a healthy eating blog

SUMMARY:
The purpose of this study is to determine if a nutrition intervention provided through a healthy eating blog is feasible and acceptable.

DETAILED DESCRIPTION:
Participants randomised to the experimental group are exposed to one blog post each week for a period of 6 months. Blog posts focus on the improvement of fruits and vegetables consumption targeting four main determinants of the behavior: (1) knowledge; (2) attitude; (3) self-efficacy; and (4) motivation/goals. Each post included a step-by-step recipe developed by the research team and featuring fruits and vegetables. Recipes were described textually and also using pictures and/or video. Twenty-six posts were created over the six-month intervention. Participants randomised to the control group are not exposed to the healthy eating blog. Feasibility (compliance, dropout and participation rates) and acceptability (satisfaction) of the study were assessed.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 and older;
* with Internet access as well as an active e-mail address;
* consuming five or less servings of F&V per day;
* living in the Quebec City metropolitan.

Exclusion Criteria:

* women dieting,
* currently pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Compliance rates | 6 months

SECONDARY OUTCOMES:
Satisfaction of the healthy eating blog intervention using Questionnaire | 6 months
  Questionnaire
Dropout rates | 6 months
Participation rates | 6 months

IPD SHARING:
Plan to Share IPD: No